CLINICAL TRIAL: NCT00556309
Title: Optical Coherence Tomography Imaging of Post Coil Aneurysm Healing.
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Marlon Mathews, M.D., Department of neurosurgery, University of California, Irvine
Other Study IDs: 20065031
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Tool: Optical Coherence Tomography Imaging of Post Coil Aneurysm Healing.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Optical Coherence Tomography Imaging of Post Coil Aneurysm Healing.
  Other Names: Optical Coherence Tomography Imaging

SUMMARY:
The purpose of this study is to identify the healing of aneurysms in three month use Optical Coherence Tomography image to measure outcomes in post coiled aneurysms. Endovascular therapeutic coiling is a widely used procedure in the management of aneurysms, which is an angiogram .

DETAILED DESCRIPTION:
Subarachnoid hemorrhage secondary to ruptured cerebral aneurysms, unruptured aneurysms that are being treated using endovascular coiling. The researcher can use Optical Coherence Tomography image at the rime of initial angiography with unruptured aneurysms, and at the three month follow up catheter angiogram.

Optical Coherence Tomography image can follow the therapeutic coiling of the aneurysm, the 6F endocatheter and the microcatheter used for the coiling procedure place in the internal carotid artery and parent artery lumen follow with Optical Coherence Tomography fiber insert through the lumen of the tube on which the image can obtain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Subject diagnosis of aneurysm and undergoing endovascular coiling

Exclusion Criteria:

* Pregnant women
* Age ≤ 18 years of age
* Patient presenting emergently with acutely ruptured aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Aneurysm Healing | up to 12 months
  Optical Coherence Tomography Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Marlon Mathew, MD, Principal Investigator — UCIMC; Zhongping Chen, PhD, Principal Investigator — Zhongping Chen, PhD, Assistant Professor, Beckman Laser Institute
Locations (2):
- United States (2):
  - Beckman Laser Institute,University of California, Irvine, Irvine, California
  - Neurosurgery department, University of California,Irvine, Irvine, California